

# Statistical Analysis Plan

# **STELLAR**

Safety and Effectiveness Evaluation of the Multi-Electrode Radiofrequency Balloon Catheter for the Treatment of Symptomatic Paroxysmal Atrial Fibrillation

Protocol# BWI\_2017\_04 (v 11.0)

Version 4.0

November 15, 2022

Sponsor: BIOSENSE WEBSTER, INC.

33 Technology Dr., Irvine, CA 92618

USA

Biosense Webster, Inc


History of Changes:

Biosense Webster, Inc



Biosense Webster, Inc






# Safety and Effectiveness Evaluation of the Multi-Electrode Radiofrequency Balloon Catheter for the Treatment of Symptomatic Paroxysmal Atrial Fibrillation (STELLAR)

**Statistical Analysis Plan Version: 4.0** 

**Corresponding to: Protocol Version: 11.0** 

The following individuals have reviewed this version of the Statistical Analysis Plan and are in agreement with the content:



Franchise Clinical Platform Lead:

Kendra McInnis Senior Director, Clinical Research

| KENDRA | Digitally signed by KENDRA MCINNIS DN: c=US, o=JNJ, ou=Subscribers, 0.9.2342.19200300.1 Page 300.1 am approving this document. Date: 2022.11.15 17:31:16 -0800' Adobe Acrobat DC version: 2015.006.30527 | 00.1.1=361800, cn=KENDRA MCINNIS |
|---|---|---|
| (Print) | (Sign) | Date |


## **List of Abbreviations**

AAD antiarrhythmic drug

AF atrial fibrillation

AFEQT Atrial Fibrillation Effect on QualiTy-of-life

AFL atrial flutter

AT atrial tachycardia

DCCV Direct Current cardioversion

DMC Data Monitoring Committee

mITT Modified Intent-To-Treat

MoCA Montreal Cognitive Assessment

NAE neurological assessment evaluable subgroup

NIHSS National Institutes of Health Stroke Scale

PAE primary adverse event

PAF paroxysmal atrial fibrillation

PP per-protocol

PV pulmonary vein

PVI pulmonary vein isolation

RF radiofrequency

SADE serious adverse device effects

SAE serious adverse event

USADE unanticipated serious adverse device effects

#### 1 STUDY DESIGN

This clinical investigation is a prospective, multicenter, single arm clinical evaluation utilizing the Biosense Webster HELIOSTAR<sup>TM</sup> catheter, in conjunction with the LassoStar<sup>TM</sup> catheter and Multi-Channel RF Generator, for the treatment of drug refractory symptomatic paroxysmal atrial fibrillation (PAF) with pre-specified performance goals for safety and effectiveness.

An adaptive Bayesian design will be used to determine the sample size. Up to a maximum of 400 evaluable subjects with symptomatic PAF may be enrolled in the main study phase.

To minimize the learning curve effect on the evaluation of safety and effectiveness of the HELIOSTAR<sup>TM</sup> catheter, a maximum of 240 roll-in subjects will be enrolled in the study. One (1) to three (3) roll-in subjects will be prospectively assigned to each ablating physician per the physician training charter. These subjects will not be counted towards the enrollment cap of 400 evaluable subjects. All subjects will be evaluated at 7 days, 1, 3, 6 and 12 months following the index procedure. Data for roll-in subjects will be analyzed separately from the main phase.

A focused neurological evaluation will be integrated within the Main Study. Forty (40) subjects enrolled in the main study will be included in the Neurological Assessment Evaluable (NAE) subset. NAE subjects will be assessed for incidence of post-ablation symptomatic and asymptomatic cerebral emboli.

Forty (40) subjects enrolled in the main study will be included in the CT/MRA subset. Subjects in the CT/MRA subset will undergo the CT/MRA exams at baseline and 3 months post ablation procedures for the assessment of PV stenosis. A subject may be permitted to participate in both the NAE and CT/MRA assessments.

### 2 TREATMENT ASSIGNMENT

This is a single-arm study. All subjects will be treated with the HELIOSTAR<sup>TM</sup> catheter.

## 3 RANDOMIZATION AND BLINDING PROCEDURES

This study is a non-randomized single-arm study. Therefore, masking of treatment assignment for operators and subjects will not be performed.

This study will employ several measures to minimize operational bias.

- Screening logs will be maintained at sites to confirm consecutive eligible subjects are considered for participation in the study
- Timing of the interim analyses for sample size selection will not be revealed to sites
- An independent statistician will be responsible for performing interim analyses

Biosense Webster, Inc

- Results from the interim analyses will not be shared with the Sponsor or sites unless the interim analysis results in a decision to stop enrollment or to file for approval
- Sponsor personnel directly involved in the conduct of the study will not have access to intermediate aggregated summaries of primary or secondary safety and effectiveness endpoint data until preparation for filing for approval

















































# 9 REFERENCES

[1] Broglio KR, Connor JT, Berry SM. (2014) Not too big, not too small: A Goldilocks approach to sample size selection. J Biopharmaceutical Statistics. 24(3):685-705.

Biosense Webster, Inc

- [2] DerSimonian R, Laird N. (1986) Meta-analysis in clinical trials. Controlled Clinical Trials 7: 177-188.
- [3] Atrial Fibrillation Effect on QualiTy-of-life (AFEQT<sup>TM</sup>) Questionnaire Instruction and Scoring Manual (2009), Version 1.0, St Jude Medical Inc.























